CLINICAL TRIAL: NCT04629326
Title: PD-L1 Targeting Molecular Imaging of Solid Tumors
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Peking University Cancer Hospital & Institute (Other)
Responsible Party: Principal Investigator, Hua Zhu, Associate Professor, Peking University Cancer Hospital & Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: WL12-Tumor
Record Dates: First submitted 2020-11-10; First posted 2020-11-16 (Actual); Last update posted 2024-08-19 (Actual); Status verified 2024-08

CONDITIONS: Gastrointestinal Tumors
MeSH Terms: conditions — Digestive System Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Imaging cohort (Experimental): All study participants will be allocated to this arm (single-arm study).Study participants will undergo 68Ga-WL12 PET/CT scans
  Interventions: Other: 68Ga-WL12 PET/CT

INTERVENTIONS:
Other: 68Ga-WL12 PET/CT — WL12, labeled with PET radio-nuclide ( Ga-68 )will be used as a molecular imaging tracer for PET/CT scanning

SUMMARY:
The objective of the study is to constrcut a noninvasive approach WL12 PET/CT to detect the PD-L1 expression of tumor lesions in patients with gastrointestinal tumors and to identify patients benefiting from anti-PD-1/L1 treatment.

ELIGIBILITY:
Inclusion Criteria:

* 1. Aged >18 years old; ECOG 0 or 1;
* 2. Patients with Gastrointestinal tumors;
* 3. Has at least one measurable target lesion according to Response Evaluation Criteria in Solid Tumors (RECIST V1.1);
* 4. life expectancy >=12 weeks.

Exclusion Criteria:

* 1. Significant hepatic or renal dysfunction;
* 2. Is pregnant or ready to pregnant;
* 3. Cannot keep their states for half an hour;
* 4. Refusal to join the clinical study;
* 5. Suffering from claustrophobia or other mental diseases;
* 6. Any other situation that researchers think it is not suitable to participate in the experiment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2021-07-20 (Actual); Primary Completion 2024-11 (Estimated); Study Completion 2024-11 (Estimated)

PRIMARY OUTCOMES:
Standardized uptake value（SUV） | 2 years
  The uptake of the tracer in the primary and metastatic tumor lesions by measuring standardized uptake value（SUV）on PET/CT

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Cancer Hospital, Beijing, Beijing Municipality, China